CLINICAL TRIAL: NCT04016649
Title: The Mechanical Characterisation of Human Saphenous and Popliteal Vein
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Collaborators: University of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Professor Eamon Kavanagh Prinicipal Investigator, University Hospital of Limerick
Other Study IDs: DVS004
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Human saphenous and popliteal vein tissue segments deemed waste following varicose vein procedures, lower limb amputation and lower limb bypass surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Non-interventional study aiming to ascertain the mechanical properties of human saphenous and popliteal vein tissue.

DETAILED DESCRIPTION:
The aim of this study is to mechanically characterise saphenous and popliteal vein segments that have been deemed waste following varicose vein procedures, lower limb amputation and lower limb bypass surgery.

By characterising the stress-stretch relationship of the vein vessel wall, treatment techniques can be better understood. Mechanical device design can be bteer informed and the the suitability of vein as a conduit for bypass and AVF procedures can be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients aged 18 years or older
* Patients undergoing varicose vein procedures or;
* Patients undergoing lower limb amputation or;
* Patients undergoing lower limb bypass surgery

Exclusion Criteria:

* Patients unable to give informed consent
* Seriously ill/unconscious patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of individuals under the care of a Vascular Consultant. Patients will be asked to participate if they are going for a procedure in which there will be vein tissue waste that would usually be discarded in the operating theatre. The procedures of interest are Varicose Vein Procedures, Lower Limb Amputation and Lower Limb Bypass Surgery.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-03-21 (Estimated)

PRIMARY OUTCOMES:
The identification of vein tissue mechanical distension and stretching properties. | 2 years
  Vein tissue will undergo inflation-extension testing and unilaxial testing. The vein tissue will be cross-sectioned and rings of venous tissue will be mechanically characterised according to the properties exhibited.

CONTACTS AND LOCATIONS:
Overall Officials: Eamon Kavanagh, MD FRCSI, Principal Investigator — University Hospital of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No
Vein Tissue will be shared with research collaborators at the Univeristy of Limerick for the purpose of mechanical characterisation.
  Patient data will not leave the site of origin. No patient identifiable data will be shared. Vein tissue sample will be labelled with a study number and dated. No patient identifiable data will be labelled on the specimen container.